CLINICAL TRIAL: NCT06000566
Title: Drug Compliance and Affecting Factors in Juvenile Idiopathic Arthritis
Status: Completed | Type: Observational
Sponsor: Yesfa Sebnem Ozbay (Other)
Responsible Party: Sponsor-Investigator, Yesfa Sebnem Ozbay, M.D., Assistant Professor, Principal investigator, Istanbul University
Organization: Istanbul University (Other)
Other Study IDs: Sponsor-Investigator
Record Dates: First submitted 2023-06-12; First posted 2023-08-21 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Arthritis, Juvenile Rheumatoid; Medication Adherence; Quality of Life
MeSH Terms: conditions — Arthritis, Juvenile; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric JIA patients: No interventions will be administered

SUMMARY:
The goal of this observational study is to learn about the drug compliance of patients with juvenile idiopathic arthritis and, to figure our factors that affect the compliance.

The main questions it aims to answer are:

* Medication use and compliance in children with chronic diseases is an important problem, but do patients with JIA really use their medications in harmony?
* Does the level of adherence to medications affect the quality of life of patients with JIA?

Participants will be asked to fill the demographic form which includes personal information and nutritional habbits, Morisky Drug Compliance Scale - 8 and the pediatric quality of life inventory forms, with attending researcher Yesfa Sebnem Ozbay, M.D.

This study is not an interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Being followed up with the diagnosis of Juvenile Idiopathic Artritis (JIA) from the pediatric rheumatology outpatient clinic of Istanbul University, Istanbul Faculty of Medicine

Exclusion Criteria:

* Refusal of patients or their parents to participate in the study
* Although the patient is followed up with the diagnosis of JIA, not using medication

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric group of age (0 to 18 years), all patients diagnosed with JIA, all patients are using drugs for their diagnose
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Drug Compliance by Morisky Medication Adherence Scale 8 (MMAS-8) | November 2022 - August 2023
  Drug adherence is a hot topic and a big issue among children and adolescents. Drug adherence among chronically ill pediatric patients will be evaluated with Morisky Medication Adherence Scale 8. With a sum of scores equalling 8, 6 to <8, or <6, patients can be categorized as having high, medium or low adherence to therapy, respectively.
Disease activation score | November 2022 - August 2023
  The activation score of the disease which will be measured by JADAS. This will help to understand the severity of the disease. JADAS consists of four items; the joint count, the physician and the patient's/parent's global assessment and the erythrocyte sedimentation rate (ESR) as an inflammatory marker. C-reactive protein (CRP) has been suggested as an alternative inflammatory marker. A higher JADAS score indicates higher disease activity as a lower JADAS score indicates lower disease activity
PedsQL (Pediatric Quality of Life Inventory) | November 2022 - August 2023
  The quality of life will be evaluated by Pediatric Quality of Life Inventory (PedsQL). Items in PedsQL are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better quality of live.
  It is aimed to evaluate the quality of life scores of juvenile idiopathic arthritis patients.

SECONDARY OUTCOMES:
Descriptice characteristics outcome measure | November 2022 - May 2023
  The correlation between the education level of the patients, nutritional habits of the patients, the socio-cultural status of the families and drug compliance is also evaluated for each patient.
Details of medication | November 2022 - May 2023
  The number of drugs used and the number of swintches between drugs will be evaluated in detail and these data will be evaluated in terms of drug compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Nuray Aktay Ayaz, M.D, M.Sci, Prof, Study Chair — IstabulU
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)